CLINICAL TRIAL: NCT02280486
Title: Efficacy and Safety of Saxagliptin and Glimepiride in Chinese Patients With Type 2 Diabetes Controlled Inadequately With Metformin Monotherapy (SPECIFY Study) : a 48-week, Multi-center, Randomized, Open-label Trial
Brief Title: Efficacy and Safety of Saxagliptin VS. Glimepiride in Chinese T2DM Patients Controlled Inadequately With Metformin
Acronym: SPECIFY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Zhongda Hospital (Other); Nanjing PLA General Hospital (Other); Changzhou No.2 People's Hospital (Other); The First Affiliated Hospital of Soochow University (Other); Wuxi People's Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Huai'an First People's Hospital (Other)
Responsible Party: Principal Investigator, Dalong Zhu, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISSSAXA0014
Record Dates: First submitted 2014-10-23; First posted 2014-10-31 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-03

CONDITIONS: Type 2 Diabetes
Keywords: saxagliptin; glimepiride; metformin monotherapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saxagliptin (Active Comparator): The treatment of saxagliptin will be initiated and maintained at 5mg every morning until the completion of the test.Meanwhile,subjects will be instructed to take stable doses of metformin (1500mg/d) through the whole trial.
  Interventions: Drug: Saxagliptin; Drug: Glimepiride
- Glimepiride (Active Comparator): Glimepiride will be initially treated with 1 mg every morning to a dose of 6 mg/day.a.m. Every 4-week the subjects will be evaluated whether reach the target fasting plasma glucose (assayed by finger-stick ≦6.1 mmol/l ). If the fasting blood glucose not achieved the target at the maximum dose, maintain the maximum dose(6mg/d) until the completion of the test.Meanwhile,subjects will be instructed to take stable doses of metformin (1500mg/d) through the whole trial.
  Interventions: Drug: Saxagliptin; Drug: Glimepiride

INTERVENTIONS:
Drug: Saxagliptin — 5 mg/d
  Other Names: Onglyza，Astrazeneca
Drug: Glimepiride — 1mg/d, up titrated 1mg if FPG >6.1 mmol/L (110mg/dL) till 6 mg
  Other Names: Amaryl，Sanofi-Aventis

SUMMARY:
This is a multi-centre, open-label, randomized, parallel trial to investigate the efficacy and safety profile of saxagliptin and glimepiride treatment in patients with type 2 diabetes inadequately controlled with metformin monotherapy.

DETAILED DESCRIPTION:
This is a multi-centre, open-label, randomized, parallel trial to investigate the efficacy and safety profile of saxagliptin and glimepiride treatment in patients with type 2 diabetes inadequately controlled with metformin monotherapy.

Screening will be made to select eligible participants before intervention. The trial will include 1-week run-in period of stable doses of metformin (1500mg) and 48-week treatment period. After the run-in period, patients were randomly assigned to one of two groups for antihyperglycaemic therapies for a total of 48-weeks: saxagliptin and glimepiride. The treatment of saxagliptin will be initiated and maintained at 5mg every morning until the completion of the study. Glimepiride will be initially treated with 1 mg every morning, and further titrated up at 4-week intervals until to reach the target fasting blood glucose (FPG).As to Glimepiride groups, if the fasting blood glucose dose not achieved the target after the maximal doses, maintain the maximal doses(6mg per day) until the completion of the study.Meanwhile, participants in both groups should take metformin 1500mg per day throughout the whole 48 weeks. At the end of the study, data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in the study subjects should fulfill the following criteria:
* Provision of informed consent prior to any study specific procedures
* Type2 diabetic patients had been on stable, maximum tolerated doses of metformin (≧1500mg/d, ≧8 weeks)
* Male or female age ≧ 25 years and ≦75 years old
* HbA1c ≧7.0 and ≦9.5%
* BMI ≧ 20 and ≦ 30 kg/m2

Exclusion Criteria:

* Subjects should not enter the study if any of the following exclusion criteria are fulfilled:
* Known or suspected allergy to trial products or related products.
* Impaired renal function defined as serum-creatinine ≥ 1.5 mg/dL (≥ 132.6 μmol/l).
* Acute or chronic disease which may cause tissue hypoxia such as cardiac or respiratory failure, shock.
* Hepatic insufficiency, acute alcohol intoxication, alcoholism.
* Subjects has a clinically significant, active (or over the past 12 months) cardiovascular history (including a history of myocardial infarction (MI), arrhythmias or conduction delays on ECG, unstable angina, or decompensated heart failure (New York Heart Association-class Ⅲ and Ⅳ).
* Proliferative retinopathy or muscular oedema requiring acute treatment.
* Lactation.
* Pregnant or positive pregnancy test at screening, nursing mother, or unwillingness to use adequate contraception (adequate contraceptive measures are sterilization, intrauterine device, oral contraceptives or barrier methods).
* Treatment with systemic corticosteroids within the past two months prior to screening.
* Tested positive for glutamic acid decarboxylase antibody.
* Receipt of any investigational drug within 1 month prior to this trial.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2015-01; Primary Completion 2016-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving glycemic response defined as Glycosylated hemoglobin (HbA1c) < 7.0% | Change from Baseline after 48 weeks treatment
  Compare the proportion of subjects after 48-week treatment achieving HbA1c<7.0%, with no hypoglycemia and no body weight gain (defined as glucose < 3.9 mmol/L with or without symptoms and weight gain < 3.0%).

SECONDARY OUTCOMES:
The change in blood glucose fluctuations of subjects. | Change from Baseline after 48 weeks treatment
  30 subjects of each group would be randomly chosen to evaluate blood glucose fluctuations by continuous glucose monitoring system (CGMS) before and after 48 weeks treatment.
The improvement in beta-cell function of subjects | Change from Baseline after 48 weeks treatment
  All subjects would be tested in fasting proinsulin, proinsulin/insulin ratio, true insulin and C-peptide during standard meal test (75-gram instant noodles) before and after 48 weeks treatment.
The change in body composition of subjects. | Change from Baseline after 48 weeks treatment
  All subjects would be measured by their weight (WT), body mass index (BMI) and waist-hip ratio (WHR) every four weeks until the end of 48 weeks treatment.
Safety and tolerability of saxagliptin vs. glimepiride measured by adverse events, serious adverse events (SAEs); laboratory assessments (biochemistry, lipids, blood and urine routine tests | Change from Baseline after 48 weeks treatment
  The proportion of AEs and SAEs would be measured.Incidence of hypoglycemia episodes (defined as symptoms with glucose < 3.1 mmol/L);adverse events (AEs);serious adverse events (SAEs);laboratory assessments (biochemistry, lipids, blood and urine routine tests);other safety and tolerability parameters (ECG, vital signs, physical examination).

CONTACTS AND LOCATIONS:
Overall Officials: Dalong Zhu, MD, PhD, Principal Investigator — the Affiliated Drum Tower Hospital of Nanjing University
Locations (1):
- at Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gu T, Ma J, Zhang Q, Zhu L, Zhang H, Xu L, Cheng J, Shi B, Li D, Shao J, Sun Z, Zhong S, Bi Y, Zhu D. Comparative effect of saxagliptin and glimepiride with a composite endpoint of adequate glycaemic control without hypoglycaemia and without weight gain in patients uncontrolled with metformin therapy: Results from the SPECIFY study, a 48-week, multi-centre, randomized, controlled trial. Diabetes Obes Metab. 2019 Apr;21(4):939-948. doi: 10.1111/dom.13605. Epub 2019 Jan 4. PMID 30520221